CLINICAL TRIAL: NCT06407856
Title: Effects of Dual Task Training on Balance and Gait in Children With Spastic Cerebral Palsy
Brief Title: Dual Task Training in Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0774
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Spastic Cerebral Palsy
Keywords: cerebral palsy; Dual-Task Training; Gait,; Balance; Cognitive-motor interference
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional therapy (Experimental): This group will only receive conventional physical therapy.
  Interventions: Other: conventional therapy
- Dual Task Training with Conventional Therapy (Experimental): This group will only receive Dual Task Training along conventional therapy
  Interventions: Other: conventional therapy; Other: Dual Task Training

INTERVENTIONS:
Other: conventional therapy — The control group embarked on a conventional therapy regimen designed for patients with spastic diplegic cerebral palsy. This group will do 10reps of ROM exercises, 3 times stretching 30sec hold with 10sec rest and 5reps of strengthening exercises, standing , weight on one leg and raising the other leg to the side or behind, putting heel in front of your toe i.e., tandem stance, standing up and sitting down from a chair without using hands, walking while alternating knee lifts with each step.This group will do conventional therapy for 30 minutes a day, 3 times a week for 8 weeks
Other: Dual Task Training — Warming up exercise Supine Trunk and lower extremity ROM exercise Main exercise Sitting Base of support: balance cushion, ball Program: perform cognition task while maintaining balance (writing, drawing, puzzle etc.) Bench sitting (half ring P.) Base of support: balance pad Program: perform fine motor activities while maintaining balance (blocks assembly, scissoring, origami etc.) Standing Base of support: balance pad, balance cushion Program: perform eating while maintaining balance (drinking water, eat a snack etc.) Cool down exercise Supine Low extremity stretching & deep breathing
  Arms: Dual Task Training with Conventional Therapy

SUMMARY:
Cerebral palsy(CP) is a non-progressive disorder, undergoing mishap to the developing brain and it affect a person's ability to move and maintain balance and posture. Old name of CP is "Little's disease". In Spastic diplegic, muscle stiffness is mainly in the legs, with the arms less affected or not affected at all. There could be secondary musculoskeletal problems due to muscle weakness resulting from poor alignment, limited range of motion, and asymmetrical posture. These deformities are negatively affected by biomechanical movements and can affect balance and gait functions. The main goal of rehabilitation in children with cerebral palsy is to restore independent walking. However, children with cerebral palsy have limited mobility, which leads to gait disorders (short steps, slow walking speed, increased swing phase and postural instability). Therefore, it is important to choose an effective training method to improve the balance and gait of children with cerebral palsy. Walking training can help improve muscle tone, postural control and gait function as well as improve muscle strength, endurance, and coordination of the lower extremities. A growing body of evidence supports implementing dual-task gait training for enhancing functional mobility and cognitive performance. This will be a randomized controlled trial, data will be collected from Rising Sun Institute, Mughalpura campus. A study will be conducted on 32 patients. Inclusion criteria of this study is spastic diplegic CP children with age between 6 to 12 years, with GMFCS level 1 to 3 and those who can walk 50 m without mechanical walking aids and maintain standing for more than 5 seconds without falling will be included. Exclusion criteria of this study is low intellectual ability (IQ < 80) and behavioral symptoms which might affect participation in the protocol, none of the children had surgery or botulinum toxin injections during the year prior to the assessment. Group1 will receive conventional therapy for 30 minutes a day, 3 times a week for 8 weeks. And group 2 will receive conventional therapy with dual-task training for 30 minutes a day, 3 times a week for 8 weeks. For the pre- and post-evaluation of all participants Berg balance scale and Gait outcome assessment list-(GOAL) will be used. Data will be analyzed through SPSS version 23.00.

ELIGIBILITY:
Inclusion Criteria:

* Participant's age will be between 6-12 years.
* Patient should be diagnosed with spastic diplegic cerebral palsy.
* GMFCS I-III

Exclusion Criteria:

* Low intellectual ability (IQ < 80) and behavioral symptoms which might affect participation in the protocol.
* If patient had any progressive neurological disorder disease.
* If he/she had surgery or botulinum toxin injections during the year prior to the assessment will also be excluded

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale | baseline and 8 weeks
  The (PBS) pediatric balance scale, a modification of the Berg Balance Scale, was developed as a balance measure for school-age children with mild-to-moderate motor impairments. It gives good test-retest and interrater reliability when used, ranged from 0.87 to 1.0
Gait Outcome Assessment List-(GOAL) | baseline and 8 weeks
  Gait Outcome Assessment List-(GOAL) is a valid assessment of gait function in ambulant children with CP. It has the potential to improve understanding of the child's and parents' priorities and thus, in conjunction with IGA, provide a more balanced assessment across the domains of theorld Health Organization's International Classification of Functioning, Disability and Health. It is a valid and reliable tool. It has a reliability of 0.92 and validity of 0.90

CONTACTS AND LOCATIONS:
Overall Officials: Tayyaba Khalid, MS*, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Yahya E, Dawes H, Smith L, Dennis A, Howells K, Cockburn J. Cognitive motor interference while walking: a systematic review and meta-analysis. Neurosci Biobehav Rev. 2011 Jan;35(3):715-28. doi: 10.1016/j.neubiorev.2010.08.008. Epub 2010 Sep 15. PMID 20833198
- [Background] Woollacott M, Shumway-Cook A. Attention and the control of posture and gait: a review of an emerging area of research. Gait Posture. 2002 Aug;16(1):1-14. doi: 10.1016/s0966-6362(01)00156-4. PMID 12127181
- [Background] Manicolo O, Grob A, Hagmann-von Arx P. Gait in Children with Attention-Deficit Hyperactivity Disorder in a Dual-Task Paradigm. Front Psychol. 2017 Jan 19;8:34. doi: 10.3389/fpsyg.2017.00034. eCollection 2017. PMID 28154547
- [Background] Carcreff L, Fluss J, Allali G, Valenza N, Aminian K, Newman CJ, Armand S. The effects of dual tasks on gait in children with cerebral palsy. Gait Posture. 2019 May;70:148-155. doi: 10.1016/j.gaitpost.2019.02.014. Epub 2019 Feb 21. PMID 30875601
- [Background] Kim GY, Han MR, Lee HG. Effect of Dual-task Rehabilitative Training on Cognitive and Motor Function of Stroke Patients. J Phys Ther Sci. 2014 Jan;26(1):1-6. doi: 10.1589/jpts.26.1. Epub 2014 Feb 6. PMID 24567664